CLINICAL TRIAL: NCT05581342
Title: Optical Coherence Tomography for Diagnosing Recurrent Basal Cell Carcinoma After Non-invasive Treatment
Brief Title: Added Value of OCT for Diagnosing Recurrent BCC After Non-invasive Treatment
Acronym: TOBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL74245.068.20
Record Dates: First submitted 2022-09-29; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Basal Cell Carcinoma
Keywords: Optical coherence tomography
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: Patients who were non-invasively treated for superficial basal cell carcinoma within five years post-treatment could be included. If CDE or OCT rose suspicion for recurrence a biopsy was obtained. When no suspicion for recurrence was raised; patients were asked to voluntarily undergo a control biopsy to verify absence of recurrence.
Who Masked: Outcomes Assessor
Masking Description: The OCT assessor was blinded to the histopathological examination of the independent dermatopathologist, whereas the dermatopathologist was blinded to the OCT assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Punch biopsy (3mm) — In case of suspicion of recurrence or a voluntary control biopsy; a punch biopsy (3mm) was obtained conform regular care.

SUMMARY:
Superficial basal cell carcinoma (sBCC) can be treated non-invasively, but follow-up is necessary because lesions can reoccur. This study aims to evaluate the additional value of optical coherence tomography (OCT) for the detection of recurrent BCC lesions, that may remain unrecognized by clinical and dermoscopic examination (CDE). This study compared the diagnostic accuracy of CDE and CDE combined with OCT for detection of recurrent basal cell carcinoma (BCC) after non-invasive treatment of sBCC.

ELIGIBILITY:
Inclusion Criteria:

* Non-invasively treated sBCC patients
* 18+ years of age

Exclusion Criteria:

* Unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
The added value of OCT for the detection of recurrent BCC | 1- 56 months post treatment
  The investigators evaluated the difference in sensitivity between CDE and CDE + OCT

SECONDARY OUTCOMES:
The number of false-positive OCT test results | 1- 56 months post treatment
  The investigators evaluated whether the addition of OCT to CDE led to false-positive test results. (i.e a decrease in specificity)
Subtyping recurrent BCC by OCT | 1- 56 months post treatment
  The investigators evaluated to what extent OCT assessors are able to correctly predict the BCC subtype of recurrent BCCs. A distinction was made between superficial BCC (sBCC; non-invasive treatment optional) and nodular/aggressive BCC (nBCC/aBCC; excision required). For BCC subtyping, sensitivity was defined as the proportion of patients with an nBCC/aBCC correctly identified by OCT as nBCC/aBCC. Specificity was defined as the proportion of patients with an sBCC correctly identified as sBCC by OCT.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limbrug, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided